CLINICAL TRIAL: NCT02998710
Title: A Multicenter, Observational, Prospective, Natural History Study of Homocystinuria Due to Cystathionine Beta-synthase Deficiency in Pediatric and Adult Patients (ACAPPELLA)
Brief Title: Natural History Study of Homocystinuria Caused by Cystathionine Beta-Synthase Deficiency (ACAPPELLA)
Status: Recruiting | Type: Observational
Sponsor: Travere Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: CBS-HCY-NHS-01
Record Dates: First submitted 2016-12-02; First posted 2016-12-20 (Estimated); Last update posted 2024-11-22 (Actual); Status verified 2024-11

CONDITIONS: Homocystinuria Due to CBS Deficiency
MeSH Terms: conditions — Homocystinuria

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of the study is to characterize the clinical course of homocystinuria in pediatric and adult patients aged 1 to 65 years under current clinical management practices

ELIGIBILITY:
Inclusion Criteria:

* Patients who are clinically diagnosed with homocystinuria
* Male/female patients aged 1 to 65 years
* Patients who consented and/or assented
* Patients who are willing and able to comply with all study-related procedures.

Exclusion Criteria:

* Medically significant postnatal complications or congenital anomalies that are not associated with homocystinuria
* Received any experimental therapy for homocystinuria during the 6 months prior to enrollment or expected to receive any such therapy during duration of the study

Ages: 1 Year to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Clinical site
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2017-01 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Changes in Met cycle metabolites levels - tHcy | 6.5 years
  Changes in total homocysteine levels in micromoles. The met cycle metabolites levels and change from baseline will be summarized using descriptive statistics at each visit.
Changes in Met cycle metabolites levels - total Cys | 6.5 years
  Changes in total cysteine levels in micromoles. The met cycle metabolites levels and change from baseline will be summarized using descriptive statistics at each visit.
Changes in Met cycle metabolites levels - Met | 6.5 years
  Changes in total methionine levels in micromoles. The met cycle metabolites levels and change from baseline will be summarized using descriptive statistics at each visit.
Changes in Met cycle metabolites levels - Cth | 6.5 years
  Changes in total cystathionine levels in micromoles. The met cycle metabolites levels and change from baseline will be summarized using descriptive statistics at each visit.
Patient Reported Outcome (PRO): Quality of Life in Neurological Disorders [Neuro-QoL] | 6.5 years
  Short forms for four domains (anxiety, depression, social activities, cognition function) by adults version for age 18+ and pediatric version for age 12-17 are used. A summary score will be calculated for each domain by adding up the scores for individual questions. The aggregated score for each domain as a continuous variable, and the change from baseline in the aggregated domain score will be summarized using descriptive statistics at each visit.
Patient Reported Outcome (PRO): Quality of Life by 36-Item Short Form Survey [SF-36] | 6.5 years
  The original responses to all questions are scored on a scale from 0 to 100, with 100 representing the highest level possible. The rescaled scores that address each specific area of functional health status are averaged together, for a final score within each of the 8 domains measured. The average is based on the number of items with non-missing scores. The average score for each domain and the change from baseline will be summarized using descriptive statistics at each visit.
National Institutes of Health (NIH) Toolbox Cognition Battery | 6.5 years
  The NIH Toolbox is a multi-dimensional assessment tool that is used to measure the neurological and behavioral function of a patient over time. Assessments are recorded as 7 individual test scores, 1 total summary score and 2 composite scores. The raw measure scores and age-corrected standard scores and the change from baseline of the scores will be summarized using descriptive statistics at each visit.
EuroQol EQ-5D™ questionnaire to measure health and quality-of-life | 6.5 years
  EQ-5D™ is a standardized questionnaire as judged by the patients. This questionnaire consists of two parts:
  1. Five domains: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension consists of 5 levels of grading: no problem, slight problem, moderate problem, severe problem and extreme problem. For youths, 3 levels of grading: no problem, some problems, and a lot of problems.
  2. Visual analogue scale (VAS) is a vertical scale from 0 (worst) to 100 (best). Descriptive statistics will be provided for the five domains. Descriptive statistics will be provided for VAS and change from baseline at each visit for pooled EQ-5D-Y version and EQ-5D-5L version.
Dual-Energy X-Ray Absorptiometry to measure bone mineral density | 6.5 years
  The z-score, t-score, and bone mineral density and change from baseline will be summarized by the location of X-ray (spine, hip, and total body) at each visit.
Eye assessments to evaluate ocular health: Visual acuity examination will be performed to determine the clarity or sharpness of vision | 6.5 years
  Visual acuity examination will be performed to determine the clarity or sharpness of vision. The results will be summarized using descriptive statistics at each visit.
Eye assessments to evaluate ocular health: Slit lamp eye examination will be performed to look for any diseases or abnormalities in the anterior portion of the eye | 6.5 years
  Slit lamp eye examination will be performed to look for any diseases or abnormalities in the anterior portion of the eye. The results will be summarized using descriptive statistics at each visit.

SECONDARY OUTCOMES:
Growth and development: World Health Organization (WHO) growth charts will be used to document height in centimeters (cm) for age 1 to 19 years old. Routine methods will be used to document height for all other age groups. | 6.5 years
  The results will be summarized using descriptive statistics at each visit.
Growth and development: World Health Organization (WHO) growth charts will be used to document Body Mass Index (BMI) in kilograms per meter square for age 1 to 19 years old. Routine methods will be used to document BMI for all other age groups. | 6.5 years
  The results will be summarized using descriptive statistics at each visit.
Growth and development: World Health Organization (WHO) growth charts will be used to document weight in kilograms (kg) for age 1 to 19 years old. Routine methods will be used to document weight for all other age groups. | 6.5 years
  The results will be summarized using descriptive statistics at each visit.
Changes in alanine aminotransferase (ALT) | 6.5 years
  The results will be summarized using descriptive statistics at each visit.
Changes in aspartate aminotransferase (AST) | 6.5 years
  The results will be summarized using descriptive statistics at each visit.
Changes in alkaline phosphatase (ALP) | 6.5 years
  The results will be summarized using descriptive statistics at each visit.
Optional homocystynuria genetic testing | The optional test will be done once at screening visit

CONTACTS AND LOCATIONS:
Overall Officials: Michael Imperiale, MD, Study Director — Travere Therapeutics, Inc.
Locations (11):
- United States (7):
  - Travere Investigational Site - Virtual Site, Culver City, California
  - Travere Investigational Site (Enrolling 1 to <5 Year-olds Only), Aurora, Colorado
  - Travere Investigational Site (Enrolling 1 to <5 Year-olds Only), Washington D.C., District of Columbia
  - Travere Investigational Site, Atlanta, Georgia
  - Travere Investigational Site, Indianapolis, Indiana
  - Travere Investigational Site, Boston, Massachusetts
  - Travere Investigational Site (Enrolling 1 to <5 Year-olds Only), Philadelphia, Pennsylvania
- Travere Investigational Site, Dublin, Ireland
- Qatar (2):
  - Travere Investigational Site, Doha, Qatar
  - Travere Investigational Site, Doha
- Travere Investigational Site, Salford, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Requests for clinical trial data, including language stating its intended use, should be directed to datarequest@travere.com. If approved, the requested information will be provided to the requestor after signing a data access agreement. Requests can be made following completion of the study and full publication of the study data in a peer reviewed journal for up to 36 months following its publication. Travere reserves the right to decline or recommend modifications to a request if it does not comply with the data sharing policy or if it is determined that the request is made by a biased source.
Time Frame: Requests can be made following completion of the study and full publication of the study data in a peer reviewed journal for up to 36 months following its publication.
Access Criteria: Requires submission and approval of intended use and a data sharing agreement.